CLINICAL TRIAL: NCT01081873
Title: A Post-Marketing Observational Study to Document Treatment Patterns and to Evaluate Leuprolide and Alternative Therapeutic Approaches to the Treatment of Advanced Prostate Cancer
Brief Title: Study to Document Treatment Patterns and to Evaluate Leuprolide and Alternative Therapeutic Approaches to the Treatments of Advanced Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PMOS-BELG-04-001
Record Dates: First submitted 2010-02-27; First posted 2010-03-05 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Prostatic Neoplasm
Keywords: Multicenter study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Advanced prostate cancer participants: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment within local reimbursement guidelines.
  Interventions: Drug: leuprolide (Lucrin/Lucrin-Tri-depot)

INTERVENTIONS:
Drug: leuprolide (Lucrin/Lucrin-Tri-depot) — Subcutaneous or intramuscular administration for all participants
  Other Names: Lucrin; Lucrin-Tri-depot

SUMMARY:
Document treatment patterns and evaluate LUCRIN / LUCRIN-TRIDEPOT® (Leuprolide) and alternative therapeutic approaches to the treatment of advanced prostate cancer during normal clinical practice and in accordance with the terms of the Belgian marketing authorization and reimbursement conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced prostate cancer who have been prescribed Lucrin/ Lucrin-Tri-depot or any other treatment with local reimbursement guidelines; Patients willing to consent to data being collected and provided to Abbott Laboratories.

Exclusion Criteria:

* Contraindications according to the Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urologists
Sampling Method: Non-Probability Sample
Enrollment: 2717 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simonne Lens, Study Director — Abbott
Locations (135):
- Belgium (131):
  - Site Reference ID/Investigator# 31147, 's-Gravenwezel
  - Site Reference ID/Investigator# 31196, Aartselaar
  - Site Reference ID/Investigator# 31237, Afsnee
  - Site Reference ID/Investigator# 31121, Alken
  - Site Reference ID/Investigator# 31170, Antwerp
  - Site Reference ID/Investigator# 31194, Antwerp
  - Site Reference ID/Investigator# 4872, Antwerp
  - Site Reference ID/Investigator# 31186, Antwerp
  - Site Reference ID/Investigator# 31141, Arlon
  - Site Reference ID/Investigator# 31199, Arlon
  - Site Reference ID/Investigator# 31247, Ath
  - Site Reference ID/Investigator# 31190, Baulers
  - Site Reference ID/Investigator# 31210, Beerse
  - Site Reference ID/Investigator# 31171, Berchem
  - Site Reference ID/Investigator# 31137, Berlaar
  - Site Reference ID/Investigator# 31204, Beveren
  - Site Reference ID/Investigator# 31184, Boutersem
  - Site Reference ID/Investigator# 31205, Braine-le-Château
  - Site Reference ID/Investigator# 31217, Brasschaat
  - Site Reference ID/Investigator# 31133, Bruges
  - Site Reference ID/Investigator# 31134, Bruges
  - Site Reference ID/Investigator# 31135, Bruges
  - Site Reference ID/Investigator# 31233, Brussels
  - Site Reference ID/Investigator# 31161, Brussels
  - Site Reference ID/Investigator# 31223, Brussels
  - Site Reference ID/Investigator# 31152, Brussels
  - Site Reference ID/Investigator# 31251, Brussels
  - Site Reference ID/Investigator# 31178, Brussels
  - Site Reference ID/Investigator# 31236, Brussels
  - Site Reference ID/Investigator# 31252, Brussels
  - Site Reference ID/Investigator# 31117, Brussels
  - Site Reference ID/Investigator# 31203, Brussels
  - Site Reference ID/Investigator# 31232, Brussels
  - Site Reference ID/Investigator# 31200, Brussels
  - Site Reference ID/Investigator# 31129, Court-Saint-Étienne
  - Site Reference ID/Investigator# 31244, Cuesmes
  - Site Reference ID/Investigator# 31208, Damme
  - Site Reference ID/Investigator# 31155, Dendermonde
  - Site Reference ID/Investigator# 31197, Dendermonde
  - Site Reference ID/Investigator# 31189, Diest
  - Site Reference ID/Investigator# 31126, Dilbeek
  - Site Reference ID/Investigator# 31116, Dworp
  - Site Reference ID/Investigator# 31160, Dworp
  - Site Reference ID/Investigator# 31179, Elingen
  - Site Reference ID/Investigator# 31249, Embourg
  - Site Reference ID/Investigator# 31166, Erpent
  - Site Reference ID/Investigator# 31192, Esneux
  - Site Reference ID/Investigator# 31188, Falmagne
  - Site Reference ID/Investigator# 31195, Feluy
  - Site Reference ID/Investigator# 31250, Floreffe
  - Site Reference ID/Investigator# 31183, Genk
  - Site Reference ID/Investigator# 31173, Genk-Waterschei
  - Site Reference ID/Investigator# 31228, Ghent
  - Site Reference ID/Investigator# 46502, Ghent
  - Site Reference ID/Investigator# 31132, Gouy-Les-Pietons
  - Site Reference ID/Investigator# 31124, Halle
  - Site Reference ID/Investigator# 31191, Hamme
  - Site Reference ID/Investigator# 31234, Hasselt
  - Site Reference ID/Investigator# 31227, Heusy
  - Site Reference ID/Investigator# 31212, Hofstade
  - Site Reference ID/Investigator# 31143, Hove
  - Site Reference ID/Investigator# 31226, Huy
  - Site Reference ID/Investigator# 31119, Izegem
  - Site Reference ID/Investigator# 31181, Izegem
  - Site Reference ID/Investigator# 31149, Knokke
  - Site Reference ID/Investigator# 31177, Koksijde
  - Site Reference ID/Investigator# 31253, Kortrijk
  - Site Reference ID/Investigator# 31130, Lasne
  - Site Reference ID/Investigator# 31159, Lennik
  - Site Reference ID/Investigator# 31123, Leper
  - Site Reference ID/Investigator# 31241, Leper
  - Site Reference ID/Investigator# 31255, Lesves
  - Site Reference ID/Investigator# 31259, Leuven
  - Site Reference ID/Investigator# 31219, Libramont
  - Site Reference ID/Investigator# 31224, Lier
  - Site Reference ID/Investigator# 31128, Liège
  - Site Reference ID/Investigator# 31144, Liège
  - Site Reference ID/Investigator# 31185, Liège
  - Site Reference ID/Investigator# 31207, Liège
  - Site Reference ID/Investigator# 31245, Liège
  - Site Reference ID/Investigator# 31243, Lommel
  - Site Reference ID/Investigator# 31225, Marcinelle
  - Site Reference ID/Investigator# 31139, Mark
  - Site Reference ID/Investigator# 31206, Mol
  - Site Reference ID/Investigator# 31153, Mons
  - Site Reference ID/Investigator# 31257, Mons
  - Site Reference ID/Investigator# 31140, Mont-sur-Marchienne
  - Site Reference ID/Investigator# 31222, Mortsel
  - Site Reference ID/Investigator# 31164, Namur
  - Site Reference ID/Investigator# 31258, Nivelles
  - Site Reference ID/Investigator# 31218, Oordegem
  - Site Reference ID/Investigator# 31156, Oosterzele
  - Site Reference ID/Investigator# 31214, Ostend
  - Site Reference ID/Investigator# 31242, Ostend
  - Site Reference ID/Investigator# 31131, Ottignies
  - Site Reference ID/Investigator# 31163, Oudenaarde
  - Site Reference ID/Investigator# 31125, Overijse
  - Site Reference ID/Investigator# 31198, Pollinkhove
  - Site Reference ID/Investigator# 31229, Ragnies
  - Site Reference ID/Investigator# 31138, Rijmenam
  - Site Reference ID/Investigator# 31122, Roeselare
  - Site Reference ID/Investigator# 31174, Roeslare
  - Site Reference ID/Investigator# 31136, Rotselaar
  - Site Reference ID/Investigator# 31180, Rumbeke
  - Site Reference ID/Investigator# 31157, Saint Truiden
  - Site Reference ID/Investigator# 31150, Saint-Denis
  - Site Reference ID/Investigator# 31215, Saint-Ghislain
  - Site Reference ID/Investigator# 31176, Saintes
  - Site Reference ID/Investigator# 31168, Schilde
  - Site Reference ID/Investigator# 31220, Schoten
  - Site Reference ID/Investigator# 31238, Schoten
  - Site Reference ID/Investigator# 31142, Seneffe
  - Site Reference ID/Investigator# 31158, Seraing
  - Site Reference ID/Investigator# 31246, Silly
  - Site Reference ID/Investigator# 31230, Sint-Genesius-Rode
  - Site Reference ID/Investigator# 31240, Sint-Niklaas
  - Site Reference ID/Investigator# 31120, Sint-Truiden
  - Site Reference ID/Investigator# 31213, Sirault
  - Site Reference ID/Investigator# 31182, Tielt
  - Site Reference ID/Investigator# 31248, Tilff
  - Site Reference ID/Investigator# 31151, Tournai
  - Site Reference ID/Investigator# 31146, Tremelo
  - Site Reference ID/Investigator# 31254, Uccle
  - Site Reference ID/Investigator# 31256, Uccle
  - Site Reference ID/Investigator# 31165, Veerle
  - Site Reference ID/Investigator# 31193, Villers-Saint-Siméon
  - Site Reference ID/Investigator# 31175, Wanze
  - Site Reference ID/Investigator# 31145, Waregem
  - Site Reference ID/Investigator# 31202, Wilrijk
  - Site Reference ID/Investigator# 31201, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe
  - Site Reference ID/Investigator# 31216, Xhendelesse
- Luxembourg (4):
  - Site Reference ID/Investigator# 31221, Bascharage
  - Site Reference ID/Investigator# 31172, Esch-sur-Alzette
  - Site Reference ID/Investigator# 31162, Ettelbruck
  - Site Reference ID/Investigator# 31231, Luxembourg

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced Prostate Cancer Participants: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines. No Baseline data was available for 3 patients who were thus excluded from all analyses.
Period: Overall Study
Arm/Group | Advanced Prostate Cancer Participants
Started | 2714 (3 patients were excluded from this and all analyses due to no available data from Baseline.)
Completed | 2416
Not Completed | 298
Not completed — Death | 86
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 142
Not completed — Progression of prostate cancer | 13
Not completed — Other | 47

BASELINE CHARACTERISTICS:
Groups:
- Advanced Prostate Cancer Participants: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines. No Baseline data was available for 3 patients who were thus excluded from all analyses. Age was available for 2,691 patients only; age was missing for 23 patients who were thus not included in the age results.
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2714
Age Continuous [Median (Full Range); unit: years] | 76.18 [46.3 to 98.2]
Age Continuous [Mean (Standard Deviation); unit: years] | 75.39 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2714

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Parameter for Staging of Prostate Cancer: Metastases at Each Visit
Description: The number of participants with metastases that are absent, local tumor, single metastases, multiple metastases in 1 organ, and multiple metastases in multiple organs at each visit is summarized.
Time Frame: time 0 (Baseline), month 3, and every 3 months until disease progression or up to 24 months, whichever came first
Population: Analysis was performed on the full analysis set (all patients for whom at least baseline data were recorded) and all available data at each visit.
Measure: Number; unit: participants
Groups:
- Advanced Prostate Cancer Participants at Baseline: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at baseline.
- Advanced Prostate Cancer Participants at Month 3: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 3.
- Advanced Prostate Cancer Participants at Month 6: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 6.
- Advanced Prostate Cancer Participants at Month 9: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had had a value recorded at Month 9.
- Advanced Prostate Cancer Participants at Month 12: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 12
- Advanced Prostate Cancer Participants at Month 15: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 15.
- Advanced Prostate Cancer Participants at Month 18: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 18.
- Advanced Prostate Cancer Participants at Month 21: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 21.
- Advanced Prostate Cancer Participants at Month 24: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a value recorded at Month 24.
- Advanced Prostate Cancer Participants - Last Available Record: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had any final value recorded.
Arm/Group | Advanced Prostate Cancer Participants at Baseline | Advanced Prostate Cancer Participants at Month 3 | Advanced Prostate Cancer Participants at Month 6 | Advanced Prostate Cancer Participants at Month 9 | Advanced Prostate Cancer Participants at Month 12 | Advanced Prostate Cancer Participants at Month 15 | Advanced Prostate Cancer Participants at Month 18 | Advanced Prostate Cancer Participants at Month 21 | Advanced Prostate Cancer Participants at Month 24 | Advanced Prostate Cancer Participants - Last Available Record
Number analyzed (Participants) | 1262 | 119 | 73 | 56 | 109 | 54 | 64 | 52 | 310 | 1411
participants
  Absent | 782 | 59 | 45 | 28 | 74 | 33 | 44 | 29 | 188 | 870
  Local tumor | 64 | 10 | 3 | 3 | 2 | 1 | 0 | 3 | 10 | 64
  Single metastases | 108 | 8 | 3 | 2 | 3 | 2 | 3 | 2 | 15 | 100
  Multiple metastases in 1 organ | 233 | 27 | 18 | 13 | 18 | 13 | 10 | 13 | 63 | 268
  Multiple metastases in multiple organs | 75 | 15 | 4 | 10 | 12 | 5 | 7 | 5 | 34 | 109

2. Primary Outcome: Effectiveness Parameter for Screening or Recurrence of Prostate Cancer: Mean Prostate-specific Antigen (PSA) at Each Visit
Description: The mean PSA in ng/mL to screen and assess for the recurrence of prostate cancer at each visit is presented.
Time Frame: time 0 (Baseline), month 3, and every 3 months until disease progression or up to 24 months, whichever came first
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Advanced Prostate Cancer Participants at Baseline | Advanced Prostate Cancer Participants at Month 3 | Advanced Prostate Cancer Participants at Month 6 | Advanced Prostate Cancer Participants at Month 9 | Advanced Prostate Cancer Participants at Month 12 | Advanced Prostate Cancer Participants at Month 15 | Advanced Prostate Cancer Participants at Month 18 | Advanced Prostate Cancer Participants at Month 21 | Advanced Prostate Cancer Participants at Month 24 | Advanced Prostate Cancer Participants - Last Available Record
Number analyzed (Participants) | 2532 | 944 | 787 | 595 | 978 | 493 | 612 | 401 | 1661 | 2595
ng/mL | 62.16 (282.64) | 12.95 (88.03) | 6.23 (34.27) | 8.01 (43.28) | 8.41 (52.84) | 8.88 (44.66) | 9.57 (57.42) | 23.02 (141.92) | 15.29 (129.06) | 30.32 (183.21)

3. Primary Outcome: Effectiveness Parameter: the Number of Participants With a Complete or Partial Response, Stable Disease, or Progressive Disease Following Treatment at Each Visit
Description: Response to treatment is summarized by the number of participants at each visit with a complete or partial response, stable disease, or progressive disease. Disease status determination was not predefined, but was based on the judgement of each Investigator.
Time Frame: month 3, and every 3 months until disease progression or up to 24 months, whichever came first
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants at Month 3 | Advanced Prostate Cancer Participants at Month 6 | Advanced Prostate Cancer Participants at Month 9 | Advanced Prostate Cancer Participants at Month 12 | Advanced Prostate Cancer Participants at Month 15 | Advanced Prostate Cancer Participants at Month 18 | Advanced Prostate Cancer Participants at Month 21 | Advanced Prostate Cancer Participants at Month 24 | Advanced Prostate Cancer Participants - Last Available Record
Number analyzed (Participants) | 1038 | 853 | 670 | 1031 | 565 | 679 | 475 | 1764 | 2210
participants
  Complete response | 525 | 496 | 402 | 668 | 347 | 401 | 276 | 1181 | 1420
  Partial response | 379 | 231 | 139 | 181 | 97 | 98 | 59 | 199 | 284
  Stable disease | 97 | 89 | 83 | 97 | 69 | 102 | 73 | 200 | 224
  Progressive disease | 37 | 37 | 46 | 85 | 52 | 78 | 67 | 184 | 282

4. Primary Outcome: Effectiveness Parameter for Prognosis: the Number of Participants With a Survival Prognosis of > 10 Years, 5 - 10 Years, 1 - 5 Years, 6 - 12 Months, and < 6 Months
Description: The prognosis for participants is summarized for each visit by the number of participants at each visit with a survival prognosis of 10 years, 5 - 10 years, 1 - 5 years, 6 - 12 months, and < 6 months. Methods for determining survival prognosis were not prespecified, but were based on the judgement of each Investigator.
Time Frame: time 0 (Baseline), month 3, and every 3 months thereafter until disease progression or up to 24 months, whichever came first
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants at Baseline | Advanced Prostate Cancer Participants at Month 3 | Advanced Prostate Cancer Participants at Month 6 | Advanced Prostate Cancer Participants at Month 9 | Advanced Prostate Cancer Participants at Month 12 | Advanced Prostate Cancer Participants at Month 15 | Advanced Prostate Cancer Participants at Month 18 | Advanced Prostate Cancer Participants at Month 21 | Advanced Prostate Cancer Participants at Month 24 | Advanced Prostate Cancer Participants - Last Available Record
Number analyzed (Participants) | 2128 | 941 | 752 | 604 | 881 | 509 | 593 | 426 | 1495 | 2365
participants
  > 10 years | 395 | 132 | 100 | 91 | 113 | 75 | 82 | 66 | 206 | 331
  5 - 10 years | 1041 | 476 | 402 | 320 | 479 | 276 | 309 | 225 | 805 | 1173
  1 - 5 years | 663 | 312 | 237 | 180 | 268 | 140 | 182 | 117 | 420 | 735
  6 - 12 months | 26 | 15 | 10 | 11 | 18 | 15 | 13 | 12 | 48 | 93
  < 6 months | 3 | 6 | 3 | 2 | 3 | 3 | 7 | 6 | 16 | 33

5. Primary Outcome: Treatment Patterns for Prostate Cancer Treatments: Number of Participants at Each Visit Who Took Lucrin/Lucrin Tridepot, Luteinizing Hormone-releasing Hormone (LHRH) Agonists, Anti-androgens, or Other Drug Treatments, or Who Had Surgery or Radiotherapy.
Description: Prostate cancer treatment for all participants is summarized by the number of participants at each visit who took any Lucrin/Lucrin Tridepot, LHRH agonist, anti-androgens, or other drug treatments, or who had any type of surgery or radiotherapy (external radiation or brachytherapy).
Time Frame: time 0 (Baseline), month 3, and every 3 months until disease progression or up to 24 months, whichever came first
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Advanced Prostate Cancer Participants - Use at Any Visit: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had used any of the treatments at any visit.
Arm/Group | Advanced Prostate Cancer Participants at Baseline | Advanced Prostate Cancer Participants at Month 3 | Advanced Prostate Cancer Participants at Month 6 | Advanced Prostate Cancer Participants at Month 9 | Advanced Prostate Cancer Participants at Month 12 | Advanced Prostate Cancer Participants at Month 15 | Advanced Prostate Cancer Participants at Month 18 | Advanced Prostate Cancer Participants at Month 21 | Advanced Prostate Cancer Participants at Month 24 | Advanced Prostate Cancer Participants - Use at Any Visit
Number analyzed (Participants) | 2714 | 1134 | 907 | 715 | 1082 | 611 | 717 | 513 | 1954 | 2714
participants
  Any Lucrin or Lucrin Tridepot used at each visit | 2028 | 1011 | 817 | 640 | 969 | 540 | 629 | 450 | 1628 | 2384
  Any LHRH agonist treatments used at each visit | 2034 | 1015 | 821 | 643 | 973 | 545 | 636 | 452 | 1635 | 2392
  Any anti-androgen treatments used at each visit | 841 | 388 | 303 | 243 | 397 | 223 | 261 | 182 | 603 | 1021
  Other drug treatments used at each visit | 31 | 22 | 21 | 24 | 31 | 27 | 24 | 23 | 57 | 86
  Any surgery performed any time up to the visit | 244 | 145 | 103 | 97 | 127 | 92 | 94 | 80 | 192 | 281
  External radiation performed any time up to visit | 129 | 84 | 76 | 73 | 79 | 43 | 56 | 33 | 133 | 228
  Brachytherapy performed any time up to the visit | 13 | 10 | 10 | 11 | 10 | 9 | 9 | 8 | 21 | 26

6. Secondary Outcome: Safety Parameter: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: The number of participants experiencing a serious adverse event during the course of the study is summarized. See the Reported Adverse Event section for details.
Time Frame: Baseline to disease progression or 24 months, whichever came first
Population: Analysis was performed on the full analysis set consisting of all patients for whom at least baseline data were recorded.
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2714
participants | 121

7. Secondary Outcome: Epidemiological Data: Mean Weight
Description: The mean weight of all participants at baseline is provided.
Time Frame: at time 0 (Baseline)
Population: Analysis was performed on the full analysis set consisting of all patients for whom at least baseline data were recorded. Data for age was available for 2,691 patients and for weight for 2,116 patients.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2714
kg | 77.36 (10.48)

8. Secondary Outcome: Epidemiological Data: Mean Age
Description: The mean age of all participants at baseline is provided.
Time Frame: at time 0 (Baseline)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2714
years | 75.39 (7.92)

9. Secondary Outcome: Epidemiological Data: Race
Description: The number of participants by race at baseline is presented.
Time Frame: at time 0 (Baseline)
Population: Analysis was performed on the full analysis set consisting of all patients for whom at least baseline data were recorded. Data for race was available for 2,217 patients.
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2217
participants
  Black | 59
  Caucasian | 2154
  Other | 4

10. Secondary Outcome: Epidemiological Data: Tumor Staging - Among Participants With a Positive Biopsy, the Number of Participants With Adenocarcinoma Tissue or Other Tissues Recorded for the Positive Biopsy.
Description: Among those participants with a positive biopsy at baseline, the number of participants with adenocarcinoma tissue or other tissue type is summarized.
Time Frame: at time 0 (Baseline)
Population: Analysis was performed on the full analysis set (all patients for whom at least baseline data were recorded) and all available data.
Measure: Number; unit: participants
Groups:
- Advanced Prostate Cancer Participants at Baseline: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines that had a tissue type recorded at Baseline.
Arm/Group | Advanced Prostate Cancer Participants at Baseline
Number analyzed (Participants) | 2279
participants
  Adenocarcinoma | 2269
  Other | 9
  Not done | 1

11. Secondary Outcome: Epidemiological Data: PSA at Baseline
Description: The median, minimum, and maximum PSA values in ng/mL at baseline are provided. The mean PSA at baseline is reported in the Primary Outcome Measure section above.
Time Frame: at time 0 (Baseline)
Population: Analysis was performed on the full analysis set consisting of all patients for whom at least baseline data were recorded. Data for PSA at baseline was available for 2,532 patients.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2532
ng/mL | 13.66 [0.0 to 6500.0]

12. Secondary Outcome: Epidemiological Data: Tumor Staging (Positive or Negative) Via a Rectal Examination, Prostate Biopsy, Echograph, or Magnetic Resonance Imaging (MRI) Test.
Description: The number of participants at baseline who were positive or negative for tumors via a rectal examination, prostate biopsy, echograph of the hyperechogenic zones, or MRI are provided.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- Advanced Prostate Cancer Participants - Rectal Examination: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines who had tumor staging assessed via rectal examination.
- Advanced Prostate Cancer Participants - Prostate Biopsy: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines who had tumor staging assessed via a prostate biopsy.
- Advanced Prostate Cancer Participants - Echograph: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines who had tumor staging assessed via an echograph (hyperechogenic zones).
- Advanced Prostate Cancer Participants - MRI: Participants with advanced prostate cancer treated with Lucrin /Lucrin- Tri-depot (leuprolide) or any other treatment with local reimbursement guidelines who had tumor staging assessed via MRI.
Arm/Group | Advanced Prostate Cancer Participants - Rectal Examination | Advanced Prostate Cancer Participants - Prostate Biopsy | Advanced Prostate Cancer Participants - Echograph | Advanced Prostate Cancer Participants - MRI
Number analyzed (Participants) | 2484 | 2364 | 2252 | 187
participants
  Positive at baseline | 2045 | 2355 | 1806 | 102
  Negative at baseline | 439 | 9 | 446 | 85

13. Secondary Outcome: Epidemiological Data: the Number of Participants With Tumor Stages T0, T1, T2, T3, and T4.
Description: The number of participants with tumor stages T0, T1, T2, T3, and T4 as reported by the physician or pathologist is summarized. T0: no evidence of primary tumor. T1: histologic tumor confined to prostate; clinically unapparent tumor, undetectable by digital rectal examination or by ultrasound. T2: tumor is confined to prostrate and can be detected by digital rectal examination. T3: tumor extends through the prostate capsule but has not spread to other organs. T4: tumor has invaded adjacent structures/organs other than seminal vesicles.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 2302
participants
  T0 stage | 30
  T1 stage | 223
  T2 stage | 614
  T3 stage | 1215
  T4 stage | 220

14. Secondary Outcome: Epidemiological Data: Node Staging - the Number of Participants With a Positive or Negative Computerized Tomography (CT) Scan or Magnetic Resonance Imaging (MRI) Test
Description: In this case, a CT or MRI is considered positive when lymph nodes are detectable. A CT or MRI is considered negative when lymph nodes are not detectable.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 1586
participants
  Positive at baseline | 374
  Negative at baseline | 1212

15. Secondary Outcome: Epidemiological Data: Node Staging - the Number of Participants With a N0 or N1 Stage at Baseline.
Description: N0: tumor cells absent from regional lymph nodes. N1: regional lymph node metastasis present.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 1656
participants
  N0 stage | 1296
  N1 stage | 360

16. Secondary Outcome: Epidemiological Data: Bone Scan at Baseline
Description: The number of participants at baseline with a positive or negative bone scan was summarized. Determination of bone scan status was based on the interpretation of the Investigator or radiologist.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 1850
participants
  Positive at baseline | 497
  Negative at baseline | 1353

17. Secondary Outcome: Epidemiological Data: Metastasis Staging (M0 or M1) at Baseline
Description: The number of participants at baseline reported to be in metastasis stage M0 or M1 is summarized. M0: no distant metastasis. M1: metastasis to distant organs beyond regional lymph nodes.
Time Frame: at time 0 (Baseline)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Advanced Prostate Cancer Participants
Number analyzed (Participants) | 1874
participants
  M0 stage | 1373
  M1 stage | 501

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported and followed to a satisfactory conclusion.
Arm/Group | Advanced Prostate Cancer Participants
Serious Adverse Events (participants affected / at risk) | 121/2714
Other Adverse Events (participants affected / at risk) | 8/2714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Prostate Cancer Participants (N=2714)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 4
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 10
Cardiac failure chronic (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 7
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Death (General disorders) | 8
Disease progression (General disorders) | 7
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 4
Multi-organ failure (General disorders) | 2
Terminal state (General disorders) | 2
Therapeutic response decreased (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Pulmonary sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Superinfection (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Cardiac enzymes increased (Investigations) | 1
Prostatic specific antigen abnormal (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diet refusal (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Bladder catheterisation (Surgical and medical procedures) | 1
Cardiac operation (Surgical and medical procedures) | 1
Angiopathy (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Infarction (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Prostate Cancer Participants (N=2714)
Porphyria non-acute (Congenital, familial and genetic disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Hot flush (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.